CLINICAL TRIAL: NCT00712673
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter 24-week Study Followed by an Extension Assessing the Efficacy and Safety of AVE0010 on Top of Metformin in Patients With Type 2 Diabetes Not Adequately Controlled With Metformin
Brief Title: GLP-1 Receptor Agonist Lixisenatide (Morning or Evening) in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Metformin
Acronym: GETGOAL-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6014; EudraCT 2007-005880-80
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia, GLP-1, metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — lixisenatide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lixisenatide (Morning Injection) (Experimental): 2-step initiation morning regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin
- Lixisenatide (Evening Injection) (Experimental): 2-step initiation evening regimen of lixisenatide: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin
- Placebo (Morning Injection) (Placebo Comparator): 2-step initiation morning regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Metformin
- Placebo (Evening Injection) (Placebo Comparator): 2-step initiation evening regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding meal (either breakfast or dinner).
  Arms: Lixisenatide (Evening Injection); Lixisenatide (Morning Injection)
Drug: Placebo — Self administered by subcutaneous injections once daily within the hour preceding meal (either breakfast or dinner).
  Arms: Placebo (Evening Injection); Placebo (Morning Injection)
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Metformin — Metformin to be continued at stable dose (at least 1.5 gram per day) up to the end of treatment.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to metformin, over a period of 24 weeks of treatment, followed by an extension.

The primary objective is to assess the effects of lixisenatide as an add-on treatment to metformin in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 24.

The secondary objectives are to assess the effect of lixisenatide, in comparison to placebo, when administered in the evening within 1 hour prior to the meal in terms of HbA1c reduction, percentage of patients reaching HbA1c less than (<) 7 percent (%), percentage of patients reaching HbA1c less than or equal to 6.5%, fasting plasma glucose (FPG), plasma glucose, plasma insulin, C-peptide, glucagon, and proinsulin during a 2-hour standardized meal test (only in morning injection arms), body weight, beta-cell function assessed by homeostasis model assessment (HOMA)-beta, fasting plasma insulin (FPI) and adiponectin; to evaluate safety, tolerability, pharmacokinetics (PK) and anti-lixisenatide antibody development, beta-cell function 4 weeks after study drug discontinuation (only in patients from the morning injection arms in some selected centers).

DETAILED DESCRIPTION:
Patients who complete the 24-week main double-blind treatment would undergo a variable double-blind extension treatment, which ends for all patients at approximately the scheduled date of Week 76 visit (Visit 25) for the last randomized patient.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit, insufficiently controlled with metformin at a stable dose of at least 1.5 gram/ day (g/day) for at least 3 months prior to screening visit

Exclusion Criteria:

* HbA1c <7% or greater than (>) 10% at screening
* At the time of screening age < legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Treatment with an antidiabetic pharmacological agent other than metformin within the 3 months preceding the screening
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* Body mass index (BMI) <=20 kilogram per square meter (kg/m^2)
* Weight change of >5 kg during the 3 months preceding the study screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis, within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening, history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting supine systolic blood pressure or diastolic blood pressure >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase: >2 times upper limit of normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); Hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody; positive serum pregnancy test in females of child bearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram, or vital signs at the time of screening that, in the judgment of the investigator or any sub-investigator, precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements [such as scheduled visits, being able to do self-injections]; likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol; investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than metformin (for example, sulfonylurea, alpha glucosidase inhibitor, other thiazolidinediones, rimonabant, exenatide, dipeptidyl-peptidase-4 inhibitors, insulin) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to study
* Any previous treatment with lixisenatide or participation in a previous study with lixisenatide
* Renal impairment defined with creatinine >1.4 mg/dL in women and creatinine >1.5 mg/dL in men
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to, gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon-like peptide-1(GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-Aventis Administrative Office, Caracas, Venezuela

REFERENCES:
- [Result] Ahren B, Leguizamo Dimas A, Miossec P, Saubadu S, Aronson R. Efficacy and safety of lixisenatide once-daily morning or evening injections in type 2 diabetes inadequately controlled on metformin (GetGoal-M). Diabetes Care. 2013 Sep;36(9):2543-50. doi: 10.2337/dc12-2006. Epub 2013 Mar 27. PMID 23536584
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Ahren B, Galstyan G, Gautier JF, Giorgino F, Gomez-Peralta F, Krebs M, Nikonova E, Stager W, Vargas-Uricoechea H. Postprandial Glucagon Reductions Correlate to Reductions in Postprandial Glucose and Glycated Hemoglobin with Lixisenatide Treatment in Type 2 Diabetes Mellitus: A Post Hoc Analysis. Diabetes Ther. 2016 Sep;7(3):583-90. doi: 10.1007/s13300-016-0179-6. Epub 2016 Jun 18. PMID 27319011
- [Derived] Yabe D, Ambos A, Cariou B, Duvnjak L, Evans M, Gonzalez-Galvez G, Lin J, Nikonova EV, de Pablos-Velasco P, Yale JF, Ahren B. Efficacy of lixisenatide in patients with type 2 diabetes: A post hoc analysis of patients with diverse beta-cell function in the GetGoal-M and GetGoal-S trials. J Diabetes Complications. 2016 Sep-Oct;30(7):1385-92. doi: 10.1016/j.jdiacomp.2016.05.018. Epub 2016 May 24. PMID 27267268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 133 centers in 16 countries between June 30, 2008 and March 09, 2011. The overall duration of treatment was at least 76 weeks (24 weeks main double-blind treatment; variable double-blind extension treatment).
Pre-assignment Details: A total of 1374 patients were screened of which 694 (50.5%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 680 patients were randomized.
Groups:
- Placebo (Morning Injection): 2-step initiation morning regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
- Placebo (Evening Injection): 2-step initiation evening regimen of volume matching placebo: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
- Lixisenatide (Morning Injection): 2-step initiation morning regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
- Lixisenatide (Evening Injection): 2-step initiation evening regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to end of treatment.
Period: Overall Study
Arm/Group | Placebo (Morning Injection) | Placebo (Evening Injection) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Started | 85 (Randomized.) | 85 | 255 | 255
Safety Population | 85 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 85 | 255 | 255
Modified Intent-to-Treat(mITT)Population | 85 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 85 | 255 | 255
Subgroup for Standardized Meal Test | 85 (Patients from morning injection arms where standardized meal test was performed.) | 0 | 255 | 0
Completed | 64 | 64 | 198 | 185
Not Completed | 21 | 21 | 57 | 70
Not completed — Adverse Event | 3 | 3 | 21 | 26
Not completed — Lack of Efficacy | 2 | 8 | 8 | 6
Not completed — Poor Compliance to Protocol | 3 | 3 | 4 | 16
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 15 | 20
Not completed — Familial and Personal Reasons | 5 | 0 | 5 | 2
Not completed — Investigator's Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo (Combined): Included all patients who received 2-step initiation morning and evening regimen of volume matching placebo.
- Total: Total of all reporting groups
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection) | Total
Number analyzed (Participants) | 170 | 255 | 255 | 680
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.4) | 54.5 (9.2) | 54.8 (10.4) | 54.7 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 89 | 157 | 141 | 387
  Male | 81 | 98 | 114 | 293
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 155 | 221 | 228 | 604
  Race: Black | 4 | 7 | 6 | 17
  Race: Asian/Oriental | 11 | 22 | 20 | 53
  Race: Other | 0 | 5 | 1 | 6
  Ethnicity: Hispanic | 49 | 96 | 98 | 243
  Ethnicity: Non Hispanic | 121 | 159 | 157 | 437
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.06 (0.90) | 8.04 (0.86) | 8.09 (0.91) | 8.06 (0.89)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 9.51 (2.28) | 9.43 (2.15) | 9.31 (2.25) | 9.40 (2.22)
2-hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — Number of patients analyzed = 169, 253 and 252 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  mmol/L | 15.51 (3.43) | 15.62 (3.97) | 15.46 (4.03) | 15.53 (3.86)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 90.15 (20.14) | 90.09 (21.10) | 89.05 (20.74) | 89.71 (20.70)
Homeostasis Model Assessment for Beta-cell Function (HOMA-beta) [Mean (Standard Deviation); unit: percentage of normal beta cells function] — Beta cell function was assessed by HOMA-beta. HOMA-beta (% of normal beta cells function) = (20 multiplied by fasting plasma insulin [micro unit per milliliter]) divided by (fasting plasma glucose [mmol/L] minus 3.5). Number of patients analyzed = 168, 251 and 252 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  percentage of normal beta cells function | 41.48 (42.12) | 42.82 (32.33) | 45.21 (46.09) | 43.38 (40.38)
Adiponectin [Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)] — Number of patients analyzed = 164, 248 and 248 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  microgram per milliliter (mcg/mL) | 5.61 (3.26) | 5.25 (2.90) | 5.25 (2.93) | 5.34 (3.01)
Fasting Plasma Insulin (FPI) [Mean (Standard Deviation); unit: picomole per liter (pmol/L)] — Number of patients analyzed = 168, 251 and 253 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  picomole per liter (pmol/L) | 75.79 (48.02) | 83.68 (63.60) | 77.90 (65.46) | 79.53 (60.84)
2-hour Postprandial Plasma Insulin (PPI) [Mean (Standard Deviation); unit: pmol/L] — Number of patients analyzed = 151, 232 and 240 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  pmol/L | 374.28 (266.55) | 380.53 (260.96) | 378.67 (328.19) | 378.30 (289.51)
Fasting C-peptide [Mean (Standard Deviation); unit: nanomole per liter (nmol/L)] — Number of patients analyzed = 164, 252 and 249 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  nanomole per liter (nmol/L) | 0.90 (0.36) | 0.97 (0.43) | 0.94 (0.43) | 0.94 (0.41)
2-hour Postprandial C-peptide [Mean (Standard Deviation); unit: nmol/L] — Number of patients analyzed = 166, 251 and 249 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  nmol/L | 2.46 (1.08) | 2.56 (1.11) | 2.42 (1.16) | 2.48 (1.12)
Fasting Glucagon [Mean (Standard Deviation); unit: nanogram per liter (ng/L)] — Number of patients analyzed = 162, 242 and 247 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  nanogram per liter (ng/L) | 87.92 (29.05) | 88.89 (32.90) | 88.53 (27.30) | 88.51 (29.88)
2-hour Postprandial Glucagon [Mean (Standard Deviation); unit: ng/L] — Number of patients analyzed = 163, 241 and 248 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  ng/L | 101.30 (33.88) | 101.46 (34.54) | 100.90 (34.12) | 101.21 (34.17)
Fasting Proinsulin [Mean (Standard Deviation); unit: pmol/L] — Number of patients analyzed = 142, 223 and 226 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  pmol/L | 31.68 (20.10) | 34.93 (24.14) | 32.35 (18.45) | 33.16 (21.16)
2-hour Postprandial Proinsulin [Mean (Standard Deviation); unit: pmol/L] — Number of patients analyzed = 139, 204 and 213 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  pmol/L | 83.48 (58.02) | 83.71 (54.65) | 77.19 (53.44) | 81.15 (55.05)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Number of patients analyzed = 168, 252 and 252 for Placebo (Combined), Lixisenatide (Morning Injection) and Lixisenatide (Evening Injection) treatment arms, respectively.
  mmol/L | 5.64 (2.81) | 6.09 (3.09) | 5.80 (3.13) | 5.87 (3.04)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 33.12 (6.45) | 33.22 (6.85) | 32.47 (5.77) | 32.91 (6.36)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 5.87 (4.72) | 6.18 (5.25) | 6.21 (5.40) | 6.11 (5.17) [0.8 to 52.1]
Duration of Metformin Treatment [Mean (Standard Deviation); unit: years] | 3.34 (3.45) | 3.73 (3.34) | 3.68 (3.90) | 3.61 (3.59)
Metformin Daily Dose [Mean (Standard Deviation); unit: milligram (mg)] | 2001.18 (439.70) | 1968.82 (446.99) | 1942.65 (406.17) | 1967.10 (430.22)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in Modified Intent-to-treat (mITT) population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Lixisenatide (Morning Injection): 2-step initiation morning regimen of lixisenatide.
- Lixisenatide (Evening Injection): 2-step initiation evening regimen of lixisenatide.
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 164 | 244 | 239
percentage of hemoglobin | -0.38 (0.075) | -0.87 (0.065) | -0.75 (0.066)
Statistical Analysis 1: Comparison: Placebo (Combined) vs Lixisenatide (Morning Injection); To detect 0.5%(or 0.4%) difference between 1 lixisenatide arm and placebo(combined), 225 patients in lixisenatide arm, 170 in placebo(combined) would provide a power of 97% (or 87%) assuming common standard deviation=1.3% with 2-sided test at 5% significance. Statistical testing:2-sided at significance level=0.05. Analysis of co-variance(ANCOVA)included treatment arms, randomization strata of screening HbA1c(<8.0,>=8.0%),BMI(<30,>=30 kg/m^2),country as fixed effects, baseline HbA1c as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Stepwise testing procedure applied to control type 1 error: lixisenatide (morning) compared with placebo (combined), if found statistically significant, then lixisenatide (evening) compared with placebo (combined); Least squares (LS) mean difference = -0.48, 95% CI 2-sided [-0.657 to -0.312], Standard Error of Mean 0.088
Statistical Analysis 2: Comparison: Placebo (Combined) vs Lixisenatide (Evening Injection); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.37, 95% CI 2-sided [-0.540 to -0.193], Standard Error of Mean 0.088

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 170 | 253 | 255
mmol/L | -0.25 (0.166) | -1.19 (0.145) | -0.81 (0.146)

3. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to the last dosing day of the study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test (patients from morning injection arms only) as pre-specified in the protocol. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- Placebo (Morning Injection): 2-step initiation morning regimen of volume matching placebo to lixisenatide.
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 64 | 200
mmol/L | -1.41 (0.588) | -5.92 (0.415)

4. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 168 | 248 | 249
kilogram | -1.64 (0.269) | -2.01 (0.234) | -2.02 (0.236)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Insulin (FPI) at Week 24
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline plasma insulin assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 157 | 237 | 229
pmol/L | -6.23 (3.254) | -5.09 (2.812) | -1.88 (2.862)

6. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Insulin (PPI) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to the last dosing day of the study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test (patients from morning injection arms only) as pre-specified in the protocol. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline PPI assessment during on-treatment period
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 54 | 181
pmol/L | -25.67 (38.028) | -87.24 (24.885)

7. Secondary Outcome: Change From Baseline in Fasting Proinsulin at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test (patients from morning injection arms only) as pre-specified in the protocol. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline proinsulin assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 48 | 154
pmol/L | -3.78 (2.246) | -7.78 (1.414)

8. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Proinsulin at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 43 | 129
pmol/L | -6.83 (5.253) | -18.88 (3.406)

9. Secondary Outcome: Change From Baseline in Fasting C-Peptide at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test (patients from morning injection arms only) as pre-specified in the protocol. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline C-peptide assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 63 | 192
nmol/L | -0.13 (0.031) | -0.10 (0.020)

10. Secondary Outcome: Change From Baseline in 2-Hour Postprandial C-Peptide at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 62 | 193
nmol/L | -0.20 (0.137) | -0.46 (0.097)

11. Other Pre Specified Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy.
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal teat. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 63 | 198
mmol/L | -0.76 (0.483) | -4.64 (0.340)

12. Secondary Outcome: Change From Baseline in Fasting Glucagon at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: Subgroup for standardized meal test (patients from morning injection arms only) as pre-specified in the protocol. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucagon assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 59 | 191
ng/L | -13.53 (3.054) | -13.27 (2.074)

13. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Glucagon at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Placebo (Morning Injection) | Lixisenatide (Morning Injection)
Number analyzed (Participants) | 62 | 191
ng/L | -12.79 (3.551) | -27.04 (2.467)

14. Secondary Outcome: Change From Baseline in Adiponectin at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline adiponectin assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mcg/mL
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 155 | 236 | 227
mcg/mL | 0.54 (0.183) | 0.55 (0.159) | 0.58 (0.160)

15. Secondary Outcome: Change From Baseline in Beta-cell Function Assessed by Homeostasis Model Assessment for Beta-cell Function (HOMA-beta) at Week 24
Description: Beta cell function was assessed by HOMA-beta. HOMA-beta (% of normal beta cells function) = (20 multiplied by fasting plasma insulin [micro unit per milliliter]) divided by (FPG [mmol/L] minus 3.5). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HOMA-beta assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: % of normal beta cells function
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 157 | 235 | 226
% of normal beta cells function | -4.16 (2.823) | 7.96 (2.450) | 4.80 (2.486)

16. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (Combined): Included all patients who received 2-step initiation, morning and evening regimen of volume matching placebo.
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 168 | 248 | 249
percentage of participants | 11.3 | 14.9 | 19.3

17. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Placebo (Morning Injection): 2-step initiation morning regimen of volume matching placebo.
- Placebo (Evening Injection): 2-step initiation evening regimen of volume matching placebo.
- Lixisenatide (Combined): Included all patients who received 2-step initiation, morning and evening regimen of lixisenatide.
Arm/Group | Placebo (Morning Injection) | Placebo (Evening Injection) | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection) | Lixisenatide (Combined)
Number analyzed (Participants) | 85 | 85 | 170 | 255 | 255 | 510
participants
  Symptomatic Hypoglycemia | 0 | 4 | 4 | 18 | 22 | 40
  Severe Symptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During the Main 24-Week Period
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 170 | 255 | 255
percentage of participants | 10.6 | 2.7 | 3.9

19. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: as for outcome 16
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 164 | 244 | 239
percentage of participants | 22.0 | 43.0 | 40.6

20. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 16
Time Frame: Week 24
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection)
Number analyzed (Participants) | 164 | 244 | 239
percentage of participants | 10.4 | 23.8 | 19.2

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration
Description: Median exposure to study treatment were 564, 561.5 and 567.5 days for the morning lixisenatide, evening lixisenatide combined placebo treatment arms, respectively.The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Lixisenatide (Combined): Included all patients who received 2-step initiation morning and evening regimen of lixisenatide.
Arm/Group | Placebo (Morning Injection) | Placebo (Evening Injection) | Placebo (Combined) | Lixisenatide (Morning Injection) | Lixisenatide (Evening Injection) | Lixisenatide (Combined)
Serious Adverse Events (participants affected / at risk) | 2/85 | 9/85 | 11/170 | 21/255 | 26/255 | 47/510
Other Adverse Events (participants affected / at risk) | 45/85 | 50/85 | 95/170 | 182/255 | 169/255 | 351/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Morning Injection) (N=85) | Placebo (Evening Injection) (N=85) | Placebo (Combined) (N=170) | Lixisenatide (Morning Injection) (N=255) | Lixisenatide (Evening Injection) (N=255) | Lixisenatide (Combined) (N=510)
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 3
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Psychosomatic disease (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 4
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Necrobiosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 1
Coronary artery bypass (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Morning Injection) (N=85) | Placebo (Evening Injection) (N=85) | Placebo (Combined) (N=170) | Lixisenatide (Morning Injection) (N=255) | Lixisenatide (Evening Injection) (N=255) | Lixisenatide (Combined) (N=510)
Bronchitis (Infections and infestations) | 8 | 6 | 14 | 22 | 6 | 28
Gastroenteritis (Infections and infestations) | 4 | 4 | 8 | 14 | 12 | 26
Influenza (Infections and infestations) | 5 | 9 | 14 | 30 | 28 | 58
Nasopharyngitis (Infections and infestations) | 11 | 15 | 26 | 38 | 20 | 58
Pharyngitis (Infections and infestations) | 2 | 3 | 5 | 6 | 16 | 22
Upper respiratory tract infection (Infections and infestations) | 6 | 10 | 16 | 22 | 15 | 37
Urinary tract infection (Infections and infestations) | 2 | 5 | 7 | 15 | 10 | 25
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 5 | 23 | 28 | 51 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 5 | 6 | 11 | 18 | 14 | 32
Headache (Nervous system disorders) | 8 | 20 | 28 | 49 | 42 | 91
Hypertension (Vascular disorders) | 3 | 6 | 9 | 17 | 15 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 7 | 10 | 9 | 19
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 4 | 14 | 6 | 20
Abdominal pain upper (Gastrointestinal disorders) | 3 | 6 | 9 | 11 | 10 | 21
Diarrhoea (Gastrointestinal disorders) | 10 | 10 | 20 | 39 | 36 | 75
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 15 | 13 | 28
Nausea (Gastrointestinal disorders) | 7 | 9 | 16 | 64 | 63 | 127
Vomiting (Gastrointestinal disorders) | 6 | 3 | 9 | 35 | 40 | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5 | 18 | 9 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 12 | 21 | 21 | 42
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 14 | 9 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 18 | 12 | 30
Fatigue (General disorders) | 3 | 2 | 5 | 14 | 9 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.